CLINICAL TRIAL: NCT00938509
Title: Ibuprofen Suppositories Administration for Fever Treatment in Infants and Children
Brief Title: Ibuprofen Suppositories Administration in Infants and Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: PROF EUGENE LEIBOVITZ, DIRECTOR, DEPARTMENT OF PEDIATRIC EMERGENCY MEDICINE, SOROKA UNIVERSITY MEDICAL CENTER
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sor477208ctil
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2009-07

CONDITIONS: Fever
Keywords: IBUPROFEN; CHILDREN; FEVER
MeSH Terms: conditions — Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: ibuprofen suppositories — 5-10 mg/kg/day-suppositories

SUMMARY:
The study will evaluate the efficacy of Ibuprofen administered as suppositories in the treatment of fever in infants and children. Ibuprofen as suppositories is not yet registered in Israel, although widely used in Europe.

DETAILED DESCRIPTION:
The drug will be used in 100 consecutive infants and children admitted with fever at the pediatric ER of the Soroka Medical Center. The information on the drug efficacy will be collected in appropriate parental questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Infants and children with rectal temperature > 38.5 C

Exclusion Criteria:

* Infants < 6 months of age

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Fever decrease | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- pediatric emergency room, SOROKA MEDICAL CENTER, Beersheba, Israel